CLINICAL TRIAL: NCT00049985
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Impact of Subcutaneous (SC) Darbepoetin Alfa Treatment on Exercise Tolerance in Subjects With Symptomatic Heart Failure (CHF) and Anemia.
Brief Title: Heart Failure and Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20010170
Record Dates: First submitted 2002-11-18; First posted 2002-11-19 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Heart Failure; Anemia
MeSH Terms: conditions — Heart Failure; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin Alfa

SUMMARY:
The purpose of this study is to determine whether increasing hemoglobin concentration in patients with heart failure and anemia will improve the patients' functional status, including exercise tolerance and New York Heart Association (NYHA) classification.

ELIGIBILITY:
Inclusion Criteria: - At least 21 years of age - Symptomatic CHF for at least 3 months - Limited exercise tolerance on a treadmill - Reduced left ventricular ejection fraction - Stable heart failure medication - Hemoglobin concentration between 9.0 and 12.5 g/dL Exclusion Criteria: - Hypertension - Unstable angina pectoris or recent myocardial infarction - Likely to receive cardiac transplant - Unable to do cardiopulmonary exercise testing - Major organ transplant (e.g., lung, liver, heart) or in renal replacement therapy (e.g., dialysis) - Recent or current treatment for malignancy - Systemic hematologic disease - Anemia due to acute or chronic bleeding - Recent epogen or darbepoetin alfa therapy - Recent blood transfusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-07

PRIMARY OUTCOMES:
Exercise tolerance

SECONDARY OUTCOMES:
NYHA classification; patient-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Ghali JK, Anand IS, Abraham WT, Fonarow GC, Greenberg B, Krum H, Massie BM, Wasserman SM, Trotman ML, Sun Y, Knusel B, Armstrong P; Study of Anemia in Heart Failure Trial (STAMINA-HeFT) Group. Randomized double-blind trial of darbepoetin alfa in patients with symptomatic heart failure and anemia. Circulation. 2008 Jan 29;117(4):526-35. doi: 10.1161/CIRCULATIONAHA.107.698514. Epub 2008 Jan 14. PMID 18195176
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com